CLINICAL TRIAL: NCT05420844
Title: Pilot Study to Evaluate the Feasibility and Acceptability of a Voice Journaling Application in Adolescents With Cystic Fibrosis
Brief Title: Pilot Study to Evaluate a Voice Journaling Application in Adolescents With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-4821
Record Dates: First submitted 2022-05-18; First posted 2022-06-15 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kintsugi (Other): Enrolled participants who will be using the Kintsugi voice journaling phone application.
  Interventions: Other: Kintsugi voice journaling application

INTERVENTIONS:
Other: Kintsugi voice journaling application — Participants will use the Kintsugi voice journaling phone application for three months.

SUMMARY:
The overall goal of this pilot study is to evaluate the feasibility and acceptability of the Kintsugi voice journaling app in adolescents with CF to inform the design of future observational and interventional trials. Additionally, the investigators aim to evaluate the potential impact of the voice journaling app on key clinical outcomes in CF.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cystic fibrosis based on sweat chloride (≥60) or two known disease-causing mutations
2. Age 14 - 18 years
3. History of elevated GAD-7 and/or PHQ-9 on screening questionnaires completed during routine CF clinical visits within the past year
4. Clinically stable at the time of enrollment, without increased respiratory and/or GI symptoms or treatment with IV and/or oral antibiotics for an acute illness for the 14 days prior to enrollment visit. Participants receiving inhaled antibiotics every other month are eligible to enroll. Participants receiving chronic oral antibiotics, including thrice weekly azithromycin will be eligible to participate
5. Access to an iOS device (iPhone or iPad) and internet/data plan
6. Parent/participant enrolled in MyChart
7. Willing to participate in study after informed consent and assent has been obtained
8. English speaking

Exclusion Criteria:

1. Endorsement of suicidal ideation on the baseline PHQ-9 (item 9) questionnaire at the enrollment visit
2. Developmental or cognitive delay preventing participant from interacting with voice journaling app
3. Unable to speak and write proficiently in English
4. Enrollment in another behavioral health study
5. Actively in treatment with a mental health provider

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Kintsugi Usage | 3 Months
  Establish the feasibility of the Kintsugi voice journaling app in participants. The investigators expect that the use of the voice journaling app will be feasible based on the frequency of use by participants over a three-month period. Frequency will be assessed on number of individual journal entries completed by participants.
Kintsugi Satisfaction | 3 Months
  Establish the acceptability of the Kintsugi voice journaling app in participants. Likert scales will be utilized in the satisfaction survey and the percentage for each answer will be reported to determine acceptability of the application. Possible responses range from "Strongly Disagree" to "Strongly Agree" with "Strongly Agree" indicating a better outcome.

SECONDARY OUTCOMES:
Change in GAD-7 (Generalized Anxiety Disorder-7) Scores | 3 Months
  The GAD-7 (Generalized Anxiety Disorder-7) scale is used for screening, diagnosis and severity assessment of anxiety disorder. Possible scores range from 0 to 21, with higher scores indicating a worse outcome.
Change in PHQ-9 (Patient Health Questionnaire-9) Scores | 3 Months
  The PHQ-9 (Patient Health Questionnaire-9 measures depression severity. Possible scores range from 0 to 27, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Hoppe, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No